CLINICAL TRIAL: NCT04985708
Title: Carolinas Cardiogenic Shock Initiative
Acronym: CCSI
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00082325; 011913E (Other: Atrium)
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2021-07

CONDITIONS: Cardiogenic Shock; Acute; Myocardial Infarction, Complications
Keywords: cardiogenic shock; Impella; shock severity index
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with AMICS are likely to benefit from MCS: later
  Interventions: Other: data collection of clinically available procedures
- Develop and maintain a patient registry of AMICS: later
  Interventions: Other: data collection of clinically available procedures
- Classify patients based on shock severity.: later
  Interventions: Other: data collection of clinically available procedures

INTERVENTIONS:
Other: data collection of clinically available procedures — when to place Impella related to PCI in patients with AMICS
  Other Names: Impella timing

SUMMARY:
To determine if deferred or delayed implantation of Impella device based on shock severity index is non-inferior with respect to 1 month and 1 year mortality compared to standard clinical protocols that do not differentiate based on shock severity in adult patients following an initial diagnosis of acute myocardial infarction complicated by cardiogenic shock (AMICS).

DETAILED DESCRIPTION:
The Carolinas Cardiogenic Shock Initiative is a clinical pathway and process improvement protocol already agreed upon by participating sites, to improve care by using a standardized algorithm to treat patients with AMI and CS. This prospective registry will capture data from this protocol as a multi-site research project in parallel with this standardized non-research clinic workflow protocol. Participating providers will follow the clinical protocol as standard of care for AMICS patients, as clinically appropriate. Patients who have been admitted and diagnosed with AMICS and meet all eligibility criteria will have their data entered in this registry.

All eligible patients who are discharged alive from the hospital will be entered into the registry and follow-up via the EMR and/or SSDI will occur at 30 days and one year to assess mortality. No additional provider appointments or further testing will be required as a part of this Registry, other than what each provider feels is medically necessary and indicated as a part of the patients' care plan.

Treatment decisions and timing will follow an approved clinical protocol and algorithm (see Appendix A) based on shock severity classification. The research team at each site will capture data generated during standard of care lab tests and clinical procedures, as well as data collected during clinical visits from eligible patients. Our target accrual is approximately 672 patients, cumulative across all participating sites.

Many of the patient specific outcomes and variables of interest for this study, are already submitted to the National Cardiovascular Data Registry (NCDR). Some additional data elements, as described in Apendix C, will also be captured. There are no benefits in participation other than the scientific knowledge gained, and the only alternative to participation is not participating.

4.1.1 Primary Outcome Variable The primary outcome variable will be 30-day all cause mortality. 4.1.2 Secondary Outcome Variable(s)

Key secondary outcome variables for analysis may include but are not limited to:

* One year mortality
* length of ICU care
* requirement for renal replacement therapy
* dose and duration of catecholamine therapy
* requirement for implantation of an active LVAD or referral for cardiac transplantation
* time to support (arrival to tertiary facility to implantation)
* use of right heart catheterization
* Attainment of TIMI III flow post reperfusion
* Attainment of Cardiac power > 0.6 watts after completion of therapy
* Reduction or elimination of vasopressors and inotropic agents.
* blood products during admission
* hemolysis requiring device discontinuation
* vascular complication requiring surgery

Study Procedures:

All inpatient data on eligible patients will come from the hospital inpatient records. Once the patient is deemed eligible, their clinical data will be entered or migrated into the research registry. Additional data will be collected at approximately one month and one year following AMICS, using the EMR and the SSDI.

The following are some of the variables which will be collected and recorded within the registry:

* Demographics
* Medical history
* Admission characteristics
* Diagnostic values
* Procedure dates and times
* Procedure characteristics
* Post-procedure information
* Discharge survival
* Survival at 1 month from AMICS
* Survival at 12 months from AMICS
* Additional Quality Metrics

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of acute myocardial infarction (AMI) with ECG and/or biomarker evidence of S-T elevation myocardial infarction (STEMI) or non-S-T elevation myocardial infarction (NSTEMI)
* Systolic blood pressure < 90mm at baseline or use of inotropes or vasopressors to maintain SBP > 90 + LVEDP > 15
* Evidence of end organ hypoperfusion
* Patient undergoes PCI

Exclusion Criteria:

* Evidence of Anoxic Brain Injury
* Unwitnessed out of hospital cardiac arrest or any cardiac arrest in which return of spontaneous circulation (ROSC) is not achieved in 30 minutes
* IABP placed prior to Impella
* Patient is already supported with an Impella
* Septic, anaphylactic, hemorrhagic, and neurologic causes of shock
* Non-ischemic causes of shock/hypotension (pulmonary embolism, pneumothorax, myocarditis, tamponade, etc.)
* Active bleeding for which mechanical circulatory support is contraindicated
* Recent major surgery for which mechanical circulatory support is contraindicated
* Mechanical complications of AMI (acute ventricular septal defect (VSD) or acute papillary muscle rupture)
* Known left ventricular thrombus for which mechanical circulatory support is contraindicated
* Mechanical aortic prosthetic valve
* Contraindication to intravenous systemic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We have no reason to assume the patients who present with AMICS, will not be representative of the demographics of the region in which the participating site(s) are located. For this reason, we will not prioritize enrollment or recruitment based on demographics. Patients who present to the cardiac catheterization lab with AMICS at participating sites, and who meet inclusion criteria, will be included in the registry upon discharge. Data will be gathered in the usual manner for clinical purposes, for patients who die during their admission. The duration of the patient's enrollment in the registry is anticipated to last 1 year from AMICS. Recording of data in the registry is anticipated to last approximately 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Survival at 30-days | 30 days
  Survival at 30 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Glen J Kowalchuk, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT04985708/Prot_000.pdf